CLINICAL TRIAL: NCT03421821
Title: Extrafascial Injection Versus Subfascial Injection of Quadratus Lumborum Block for Postoperative Analgesia in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: The Difference Between the Extrafascial Injection and the Subfascial Injection of Quadratus Lumborum Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Wenquan He, Attending physician of anesthesiology department, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MZK-HWQ1
Record Dates: First submitted 2018-01-22; First posted 2018-02-05 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Postoperative Pain
Keywords: quadratus lumborum block; anterior thoracolumbar fascia; subfascial injection; extrafascial injection
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: The investigators random divided subjects into two groups, the "subfascial injection group"and the "extrafascial injection group". Two groups were injected 0.33% ropivacaine 30 ml to the target location.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Subfascial Injection Group (Experimental): 30 ml of 0.33% ropivacaine was injected to subfascial.
  Interventions: Drug: Ropivacaine
- Extrafascial Injection Group (Active Comparator): 30 ml of 0.33% ropivacaine was injected to extrafascial.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — Subfascial injection OR extrafascial injection
  Other Names: Naropin

SUMMARY:
Quadratus lumborum block can be used for the hip surgery and abdominal surgery postoperative analgesia. But the lower thoracic to the hip dermatome can't be blocked at the same time. The anesthetists used the same method, but had produced the different dermatome were blocked. The investigators hypothesized that this was due to local anesthetics was injected to different locations of the anterior thoracolumbar fascia. If the investigators inject local anesthetics to the anterior layer of thoracolumbar extrafascial, this produced the dermatomal coverage from lower abdominal to hip. A different situation was when the investigators injected local anesthetics to anterior thoracolumbar subfascia, the lower thoracic dermatome were blocked.

DETAILED DESCRIPTION:
Quadratus lumborum block can be used for the hip surgery and abdominal surgery postoperative analgesia. But the lower thoracic to the hip dermatomes can't be blocked at the same time. The anesthetists used the same method, but had produced the different dermatomes were blocked. The investigators hypothesized that this was due to local anesthetics was injected to different locations of the anterior thoracolumbar fascia. If the investigators inject local anesthetics to the anterior thoracolumbar extrafascial (between the anterior layer of thoracolumbar fascia and psoas major muscle), this produced the dermatomal coverage from lower abdominal to hip. In this case, the investigators speculated the local anesthetic spread to the lumbar paravertebral space via the fascia and the fascicle of psoas major. A different situation was when the investigators injected local anesthetics to anterior thoracolumbar subfascial (between the anterior layer of thoracolumbar fascia and quadratus lumborum), the lower thoracic dermatomes were blocked. The investigators speculate that the local anesthetic injected subfascial could spread cephalad to lower thoracic paravertebral space posterior to the endothoracic fascia via lateral arcuate ligament.

The investigators confirm the hypothesis in the pilot trial. therefore, the investigators need to trial with large sample. The investigators plan to improve the clinical guidance of quadratus lumborum block technology, so that more patients benefit.

ELIGIBILITY:
Inclusion Criteria:

* Participants undergoing laparoscopic cholecystectomy. ASA: I~II. BMI: 17~32. The operation time is less than 2 hours. Participants volunteered for the trial.

Exclusion Criteria:

* Pregnant and lactation women. Coagulation disorders. Drug allergy. Can not communicate normally. Bacteremia. Emergency surgery. ASA: >III.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-02-25 (Actual); Primary Completion 2018-09-17 (Actual); Study Completion 2018-09-17 (Actual)

PRIMARY OUTCOMES:
Changes of pain intensity of the 3 holes at 48 hours post-operation | 48 hours after operation
  The three holes include the Subxiphoid hole, Subcostal hole and supraumbilical hole in the laparoscopic cholecystectomy. Patients reported pain intensity of each hole in the post-operation of 1 hour, 6 hours, 12 hours, 24 hours, 36 hours and 48 hours. Each item is scored 0-10 (0 = no pain; 10= pain as bad as can be).

SECONDARY OUTCOMES:
Adverse effects | 48 hours after operation
  Included the Postoperative nausea and vomiting (PONV),pruritus, gastroduodenal ulcer and local anaesthetics toxicity.
Limbs weakness | at 30 min after block
  Record according to the modified Lovett rating scale (LRS). It was defined as follows: 0 = complete paralysis; 1 = almost complete paralysis; 2 = pronounced mobility impairment; 3 = slightly impaired mobility; 4 = pronounced reduction of muscular force; 5 = slightly reduced muscular force; 6 = normal muscular force.
Postoperative analgesic consumption | 48 hours after operation
  The observer recorded the consumption of parecoxib sodium and fentanyl and the point of administered time within 48 hours after operation
dependent ambulation | at 1 and 6 hours after surgery
  The proportion of dependent ambulation assistance at 1 and 6 hours after surgery in the two groups.
Sensory block level | 30 min after blocked
  The sensory level was assessed with cold sensation (ice cube) in each dermatomal distribution from T4 to L5 every 5 minutes for 4 times.
patients satisfaction | 48 hours after operation
  Patient satisfaction was assessed using a scale of 0-10, 10 being the most satisfied, at postoperative 48 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Kaizhi Lu, MD, Study Director — First affiliation hospital of third military medical university
Locations (1):
- First affiliated hospital of third military medical university, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participants data for all primary and secondary outcome measure will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel. Requestors will be required to sign a data access agreement.

REFERENCES:
- [Result] Blanco R, Ansari T, Girgis E. Quadratus lumborum block for postoperative pain after caesarean section: A randomised controlled trial. Eur J Anaesthesiol. 2015 Nov;32(11):812-8. doi: 10.1097/EJA.0000000000000299. PMID 26225500
- [Result] Ishio J, Komasawa N, Kido H, Minami T. Evaluation of ultrasound-guided posterior quadratus lumborum block for postoperative analgesia after laparoscopic gynecologic surgery. J Clin Anesth. 2017 Sep;41:1-4. doi: 10.1016/j.jclinane.2017.05.015. Epub 2017 Jun 1. PMID 28802593
- [Result] Kumar A, Sadeghi N, Wahal C, Gadsden J, Grant SA. Quadratus Lumborum Spares Paravertebral Space in Fresh Cadaver Injection. Anesth Analg. 2017 Aug;125(2):708-709. doi: 10.1213/ANE.0000000000002245. No abstract available. PMID 28654429
- [Result] La Colla L, Ben-David B, Merman R. Quadratus Lumborum Block as an Alternative to Lumbar Plexus Block for Hip Surgery: A Report of 2 Cases. A A Case Rep. 2017 Jan 1;8(1):4-6. doi: 10.1213/XAA.0000000000000406. PMID 28036319
- [Result] Wikner M. Unexpected motor weakness following quadratus lumborum block for gynaecological laparoscopy. Anaesthesia. 2017 Feb;72(2):230-232. doi: 10.1111/anae.13754. Epub 2016 Nov 28. PMID 27891579